CLINICAL TRIAL: NCT01702415
Title: Randomised, Double Blind, Placebo Controlled Trial to Ascertain the Efficacy and Safety of Intravenous Zoledronic Acid in Adult Patients With Cystic Fibrosis.
Brief Title: Zoledronic Acid in Cystic Fibrosis
Acronym: IZAC
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: Papworth Hospital NHS Foundation Trust (Other Government)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P01612
Record Dates: First submitted 2012-10-04; First posted 2012-10-08 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Cystic Fibrosis
Keywords: Cystic fibrosis; Bone density
MeSH Terms: conditions — Cystic Fibrosis | interventions — Zoledronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- Zoledronic acid (Experimental): Active IMP
  Interventions: Drug: Zoledronic acid

INTERVENTIONS:
Drug: Zoledronic acid — Single dose, intravenous solution 5mg
  Arms: Zoledronic acid
Drug: Placebo
  Arms: Placebo

SUMMARY:
Null hypotheses: zoledronic acid does not improve bone density in cystic fibrosis.

Low bone mineral density (osteoporosis) is prevalent in adults with cystic fibrosis (CF); they have an increased rate of bone fractures in comparison to the general population. CF patients start to lose bone density in adolescence/early adulthood due to an imbalance in bone breakdown and formation. Predicted survival for patients with CF has increased from 16 years in 1970 to 36.5 years in 2009 which has resulted in an increase in comorbidities associated with increased longevity in CF e.g. decreased bone density. Oral and intravenous bisphophosphonates are known to increase bone density in CF; the current licensed oral preparations require daily or weekly dosing which are difficult to maintain. Zoledronate, which is licensed for use, is administered intravenously once a year which should be easier to administer. The current evidence relates to its use in other disease groups e.g. glucocorticoid induced osteoporosis and oncology. The purpose of this study is to ascertain its efficacy in cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis
* Aged at least 18 years
* Bone mineral density score of -1.5 or less at lumbar spine or total hip
* Able to give informed consent

Exclusion Criteria:

* Previous solid organ transplant
* on solid organ transplant waiting list
* Long trem oral glucocorticosteroids
* CRP >20mg on day of randomisation
* Hypocalcaemia
* Poor dental hygiene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Bone density | 12 months
  Bone density measure by DEXA

SECONDARY OUTCOMES:
Effect of zoledronic acid on the number of bone fractures | 12 months
  Bone fractures

OTHER OUTCOMES:
Bone pain | 12 months
  Frequency and severity of bone pain as a possible side effect of zoledronic acid

CONTACTS AND LOCATIONS:
Overall Officials: Charles Dr Haworth, FRCP, Principal Investigator — Papworth Hospital NHS Foundation Trust
Locations (1):
- Papworth Hospital NHS Foundation Trust, Cambridge, Cambridgeshire, United Kingdom

REFERENCES:
- [Derived] Jeffery TC, Chang AB, Conwell LS. Bisphosphonates for osteoporosis in people with cystic fibrosis. Cochrane Database Syst Rev. 2023 Jan 10;1(1):CD002010. doi: 10.1002/14651858.CD002010.pub5. PMID 36625789